CLINICAL TRIAL: NCT02039089
Title: A Two-Part, Randomized, Double-Blind, Placebo-Controlled, Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2006 in Healthy Japanese and White Subjects
Brief Title: A Two-Part Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of E2006 in Healthy Japanese and White Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2006-A001-003
Record Dates: First submitted 2014-01-10; First posted 2014-01-17 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Part A: dose escalation of E2006 in Japanese subjects from 2.5 mg (1 x 2.5-mg tablet) up to 10 mg (1 x 10-mg tablet) then to 25 mg (2 x 10-mg tablet, 1 x 5-mg tablet).
  Interventions: Drug: E2006 2.5 mg; Drug: E2006 10 mg; Drug: E2006 25 mg
- 2 (Experimental): Part B: E2006 10 mg for White subjects that will be group matched to the Japanese subjects in the 10 mg period in Part A.
  Interventions: Drug: E2006 10 mg
- 3 (Placebo Comparator): E2006-matched placebo tablets
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2006 2.5 mg
  Arms: 1
Drug: E2006 10 mg
  Arms: 1; 2
Drug: E2006 25 mg
  Arms: 1
Drug: Placebo
  Arms: 3

SUMMARY:
This study will be a single-center, multiple-dose, randomized, double-blind, placebo-controlled, parallel-group study in healthy male and female subjects. The study will consist of 2 parts: Part A (3 cohorts of healthy Japanese subjects dosed in the evening) and Part B (one cohort of healthy white subjects dosed in the evening). The cohorts will be conducted sequentially. Part A will be started first with the 2.5-mg dose cohort, followed by the 10-mg dose cohort and then the 25-mg dose cohort. Part B will be conducted in parallel with the 10-mg cohort of Part A, with the possibility of overlap.

ELIGIBILITY:
Inclusion Criteria

Subjects have to meet all of the following criteria to be included into this study:

1. Non-smoking, male or female subjects age greater than or equal to 20 years and less than or equal to 55 years old at the time of informed consent.
2. Japanese subjects must have been born in Japan of Japanese parents and Japanese grandparents, must have lived no more than 5 years outside of Japan, and must not have changed their life style or habits, including diet, while living outside of Japan.
3. Who report habitual time in bed greater than 7 hours, with lights-out 21:00 to 24:00 hours and lights-on 06:00 to 09:00 hours.
4. Who report typical sleep latency of less than or equal to 30 minutes.
5. With typical total sleep time greater than or equal to 420 minutes.
6. Body mass index (BMI) greater than or equal to 18 and less than or equal to 28 kg/m2 at Screening.

Exclusion Criteria

Subjects who meet any of the following criteria will be excluded from this study:

1. Clinically significant illness that requires medical treatment within 8 weeks or a clinically significant infection that requires medical treatment within 4 weeks of dosing.
2. Any subject that has a known history of malaria or has traveled to a country with known malarial risk (ie, countries designated as 'high' or 'moderate' risk according to the list available at http://www.cdc.gov/malaria) within the last year.
3. Evidence of disease that may influence the outcome of the study within 4 weeks before dosing (eg, psychiatric disorders, disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism).
4. Any history of abdominal surgery that may affect PK profiles of E2006 (eg, hepatectomy, nephrotomy, digestive organ resection).
5. Any clinically abnormal symptom or organ impairment found by medical history, physical examination, vital sign and, ECG assessments, or laboratory test results that requires medical treatment.
6. A QTcF interval greater than 450 ms demonstrated on a repeated ECGs (repeated if initial ECG indicates QT greater than 450 ms) at Screening or Baseline.
7. A history or a family history of congenital QT prolongation or with a history of risk factors for torsade de pointes (eg, heart failure, hypokalemia, family history of long QT Syndrome), or use of concomitant medications that prolong the QT/QTc interval.
8. Any suicidal ideation with intent with or without a plan at Baseline or within 6 months of Baseline (ie, answering "Yes" to questions 4 or 5 on the Suicidal Ideation Section of the C-SSRS).
9. Any lifetime suicidal behavior (per the Suicidal Behavior Section of the C-SSRS).
10. Known history of clinically significant drug allergy at screening.
11. Known history of food allergies or presently (at Screening or Baseline) experiencing significant seasonal or perennial allergy.
12. Active viral hepatitis (A, B or C) as demonstrated by positive serology at Screening. Subjects with HIV infection as confirmed verbally.
13. History of drug or alcohol dependency or abuse within the 2 years before Screening, or those who have a positive urine drug test or breath (or urine) alcohol test at Screening or Baseline.
14. Habitually consumes more than 400 mg caffeine per day. Caffeine consumption must be discontinued for at least 24 hours before Baseline check-in.
15. Intake of nutritional supplements, juice, and herbal preparations or other foods or beverages that may affect the various drug metabolizing enzymes and transporters (eg, alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice, vegetables from the mustard green family [eg, kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard], charbroiled meats) within 1 week before dosing.
16. Intake of herbal preparations containing St. John's Wort within 4 weeks before dosing.
17. Use of prescription drugs within 4 weeks before dosing.
18. Intake of over-the-counter medications within 2 weeks before dosing.
19. Currently enrolled in another clinical study or used any investigational drug or device within 30 days preceding initial dose of study drug.
20. Receipt of blood products within 4 weeks, donation of blood within 8 weeks, or donation of plasma within 1 week of dosing.
21. Engagement in strenuous exercise within 2 weeks before Screening and check-in (eg, marathon running, weight lifting).
22. Diagnosis of a sleep disorder (eg, insomnia, obstructive sleep apnea, restless leg syndrome, Periodic Limb movements in Sleep, narcolepsy, circadian rhythm disorder).
23. Performed shift work within 2 weeks before Screening.
24. Had taken an airline flight across 3 or more time zones in the 7 days before Screening.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) profiles of E2006 | Up to 49 days
  The primary PK parameters are Cmax, tmax, AUC(0-T), AUC(0-24h), and t1/2, derived by non-compartmental analyses using the plasma concentration of E2006 and metabolites (as data permit).
Pharmacodynamic (PD) profile of E2006 | Up to 49 days
  acute effects of E2006 on sleepiness in the hour before bedtime as well as next-day residual sleepiness throughout the daytime hours subsequent to each dose using the KSS and PVT. Effects of E2006 on nighttime sleep will be evaluated using PSG. High-precision QT analyses (HPQT) will be performed using data from 24-hour Holter recordings. The time points of Holter readings will be corresponding to the PK time points.
Adverse events (AEs ) as a measure of safety and tolerability | Up to 49 days
Suicidality as a measure of safety and tolerability | Up to 49 days
  Measured by the columbia suicide severity rating scale (C-SSRS)
Vital signs as a measure of safety and tolerability | Up to 49 days
  Vital sign measurements will include systolic and diastolic blood pressure (BP) and pulse rate
Electrocardiogram (ECG) as a measure of safety and tolerability | Up to 49 days
  Twelve-lead ECGs will be obtained as a measure of safety and tolerability
Laboratory assessments as a measure of safety and tolerability | Up to 49 days

CONTACTS AND LOCATIONS:
Locations (1):
- Glendale, California, United States